CLINICAL TRIAL: NCT05154721
Title: Effect of Music and Rhythm Training Delivered Through a Serious Game on the Reading Skills of Children With a Specific Learning Disorder Impacting Reading, a Multicentric Double-blind and Placebo-controlled Study (Mila-Learn-01)
Brief Title: Rhythm Training of a Serious Game on the Reading Skills of Children w/ a Specific Learning Disorder Impacting Reading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poppins (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mila-Learn-01; 2021-A01709-32 (Other: French Study Registration number)
Record Dates: First submitted 2021-11-23; First posted 2021-12-13 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Learning Disorder, Specific; Learning Disabilities; Dyslexia; Specific Learning Disorder, With Impairment in Reading
MeSH Terms: conditions — Specific Learning Disorder; Learning Disabilities; Dyslexia

STUDY DESIGN:
Intervention Model Description: The experimental arm (EXPE Group) will receive the Mila-Learn game and the control arm (CONT Group) will receive the Mila-Placebo game.
  In each group, the children will follow the same training protocol consisting of five training sessions per week on the game corresponding to their group. Each game comprises 8 tasks to be completed on a touchscreen tablet. Each session lasts 25 minutes (±20%).
Who Masked: Participant, Investigator
Masking Description: In order to maintain the blinding of the patient and his/her family, the study will be presented to them as evaluating the effect of serious games on a child's learning without explaining that the study is specifically interested in the Mila-Learn game, music and rhythm.
  Evaluations will be carried out in a double-blind manner. The evaluators will not know to which group the children belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPE Group (Experimental): The experimental group (EXPE Group) will receive the Mila-Learn game.
  Interventions: Device: experimental Group - Mila-Learn
- CONT Group (Placebo Comparator): The control group (CONT Group) will receive the Mila-Placebo game.
  Interventions: Device: control Group - Mila-Placebo

INTERVENTIONS:
Device: experimental Group - Mila-Learn — Eight tasks are used in Mila-Learn.
  Arms: EXPE Group
Device: control Group - Mila-Placebo — Eight tasks similar to Mila-Learn are used in the placebo group
  Arms: CONT Group

SUMMARY:
Mila-Learn-01 is a double-blind clinical study (meaning that neither the patient nor the doctor or his/her team will know which game the child has), which enables us to see the effect of a serious game on the child's reading skills.

The patients who will participate in this research will receive, at random, one of the two serious study games, the experimental game (Mila-Learn) or the placebo game (Mila-Placebo). The tasks designed in the placebo game mirror those of Mila-Learn.

Each game comprises eight tasks to be completed on a touchscreen tablet. Each session lasts 25 minutes (±20%); five training sessions lasting 25 minutes are planned per week for eight weeks.

DETAILED DESCRIPTION:
The study consists of a randomised, double-blind clinical trial with a control group to evaluate the impact of the Mila-Learn game on children's skills. In order to maintain the blinding of the patient and his/her family, the study will be presented to them as evaluating the effect of serious games on a child's learning without explaining that the study is specifically interested in the Mila-Learn game, music and rhythm.

Each child included in the study will be randomised:

* either to the experimental group (EXPE Group) and in this case will receive the Mila-Learn game
* or to the control group (CONT Group) and will receive the Mila-Placebo game.

A randomisation list will be edited by the statistician. It will allow us to know whether the patient will be in the experimental arm or the control arm when sending out the tablets, depending on the chronological order of the inclusions, so that we can send the corresponding tablet to the patient.

In each group, the children will follow the same training protocol consisting of five training sessions per week on the game corresponding to their group. Each game comprises 8 tasks to be completed on a touchscreen tablet. Each session lasts 25 minutes (±20%).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Specific Learning Disorder with Impairment in Reading through speech therapy testing and confirmed by a doctor. Specific Learning Disorder with Impairment in Reading is defined in the diagnostic and statistical manual of mental disorders (DSM-5).
* Patient 7-11 years old, schooled from the second year of primary school (CE1) to the last year of primary school (CM2).
* Native Speaker of French OR French bilingualism at home AND Child schooled in France for more than 3 years
* Person affiliated with a social security scheme.
* Participant's agreement to participate and the agreement of the holders of parental authority and commitment to follow the protocol.

Exclusion Criteria:

* Patient undergoing or having undergone speech therapy or psychomotor therapy during the 12 months before the start of the study.
* Patient who has previously used Mila-Learn.
* Uncontrolled, chronic illness, at the investigator's discretion.
* Participation in another interventional study that could impact the analysis of the study.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of musical and rhythmic training measured by the number of pseudo-words correctly read | 8 weeks after the start of training (T2)
  Absolute change in the number of pseudo-words correctly read by the children in the pseudo-word reading test, EVALEO 6-15, by Launay, Maeder, Roustit and Touzin, 2018.

SECONDARY OUTCOMES:
Safety criteria | During the training phase, up to 8 weeks
  Descriptive evaluation of any adverse events reported by the users.
Evaluation of phonological skills measured by the Battery of Analytical Test on Written Language (BALE) initial or final phoneme deletion test | 8 weeks after the start of training (T2)
  This endpoint relates to the child's phonological skills at T2 compared to T1, evaluated using the BALE [Battery of Analytical Tests on Written Language] initial or final phoneme deletion test.
Evaluation of speed and accuracy skills by the percentage of words correctly read in two minutes | 8 weeks after the start of training (T2)
  This endpoint relates to reading skills in terms of speed and accuracy. The analysis will focus on the percentage of words correctly read in two minutes (EVAL2M, Evaleo 6-15).
Evaluation of grapheme conversion skills in terms of speed and accuracy measured by two pseudo-word transcription tests | 8 weeks after the start of training (T2)
  This endpoint relates to phoneme-grapheme correspondence skills, evaluated using two pseudo-word transcription tests.
Evaluation of self-esteem measured by the Rosenberg Self-Esteem scale ; using a 4-point scale format ranging from strongly agree to strongly disagree | 8 weeks after the start of training (T2)
  This endpoint relates to the evolution of the child's self-esteem measured by the Rosenberg Self-Esteem scale.
Evaluation of the reading skills by the children in the pseudo-word reading test, EVALEO 6-15 | 16 weeks after the start of training (T3)
  The primary endpoint is the absolute change in the number of pseudo-words correctly read by the children in the pseudo-word reading test, EVALEO 6-15, by Launay, Maeder, Roustit and Touzin, 2018.

CONTACTS AND LOCATIONS:
Overall Officials: David COHEN, Dr, Principal Investigator — Hôpital Pitié-Salpêtrière
Locations (3):
- France (3):
  - Centre médical pluridisciplinaire CogCharonne, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Centre Hospitalier Henri Laborit, Poitiers

REFERENCES:
- [Derived] Descamps M, Grossard C, Pellerin H, Lechevalier C, Xavier J, Matos J, Vonthron F, Grosmaitre C, Habib M, Falissard B, Cohen D. Rhythm training improves word-reading in children with dyslexia. Sci Rep. 2025 May 21;15(1):17631. doi: 10.1038/s41598-025-02485-y. PMID 40399331